CLINICAL TRIAL: NCT01209026
Title: A Randomised, Placebo-controlled, Four-way Crossover Repeat Dose Study to Evaluate the Effect of the Inhaled Fluticasone Furoate (FF)/GW642444M Combination on Electrocardiographic Parameters, With Moxifloxacin as a Positive Control, in Healthy Subjects
Brief Title: Corrected QT (QTc) Study With Flucticasone Furoate and GW642444
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 102936
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Asthma
Keywords: Fluticasone furoate (GW685698); moxifloxacin; QTc; GW642444; pharmacokinetics
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- FF/GW642444M (200/25mcg) (Experimental): Inhaled fluticasone furoate (200mcg) /GW642444M (25mcg) combination Days 1- 7; placebo tablet taken orally single dose (po SD) on Day 7.
  Interventions: Drug: Fluticasone furoate (200 mcg)/GW642444 (25mcg) combination; Drug: Placebo Inhaler; Drug: Moxifloxacin placebo
- FF/GW642444M (800/100 mcg) (Experimental): Inhaled fluticasone furoate (800mcg) /GW642444M (100mcg) combination Days 1- 7; placebo tablet (po SD) on Day 7.
  Interventions: Drug: Fluticasone furoate (400 mcg)/GW642444 (50mcg) combination; Drug: Moxifloxacin placebo
- Moxifloxacin (Active Comparator): Inhaled placebo on Days 1-7; moxifloxacin (400mg po SD) on Day 7
  Interventions: Drug: Placebo Inhaler; Drug: Moxifloxacin 400mg
- Placebo (Placebo Comparator): Inhaled placebo on Days 1-7; placebo tablet (po SD) on Day 7.
  Interventions: Drug: Placebo Inhaler; Drug: Moxifloxacin placebo

INTERVENTIONS:
Drug: Fluticasone furoate (200 mcg)/GW642444 (25mcg) combination — Novel dry powder inhaler
  Arms: FF/GW642444M (200/25mcg)
Drug: Fluticasone furoate (400 mcg)/GW642444 (50mcg) combination — Novel dry powder inhaler
  Arms: FF/GW642444M (800/100 mcg)
Drug: Placebo Inhaler — Matching placebo Novel dry powder inhaler. Lactose monohydrate and magnesium stearate.
  Arms: FF/GW642444M (200/25mcg); Moxifloxacin; Placebo
Drug: Moxifloxacin 400mg — Film coated oral tablet
  Arms: Moxifloxacin
Drug: Moxifloxacin placebo — Film coated oral tablet
  Arms: FF/GW642444M (200/25mcg); FF/GW642444M (800/100 mcg); Placebo

SUMMARY:
A randomised, placebo controlled thorough QTc study to evaluate the effect of repeat dose FF/GW642444M combination, with moxifloxacin as a positive control, on the QTc interval in healthy male and female subjects. Key assessments will include 12- lead electrocardiogram (ECG) and pharmacokinetic (PK) parameters, along with safety being assessed by blood pressure, heart rate, clinical laboratory safety tests, and collection of adverse events.

DETAILED DESCRIPTION:
This is a randomised, placebo controlled, four way crossover thorough QT study to evaluate the effect of repeat dose fluticasone furoate/GW642444M combination on the QTc interval in healthy male and female subjects. Up to 85 subjects will receive inhaled placebo and inhaled fluticasone furoate/GW642444M combination (200/25 microgram (mcg) or 800/100 mcg) and oral moxifloxacin (400 milligram (mg)). The inhaled treatments will be given double-blind once daily in the morning for 7 days with a single-blind placebo tablet also administered on Day 7. Moxifloxacin (positive control) will be given as a single-blind single dose on Day 7 in the morning with inhaled double-blind placebo administered in the morning on Days 1-7. Individual time-matched changes from baseline in QT duration corrected for heart rate by Fredericia's formula (QTcF) (difference from placebo) for fluticasone furoate/GW642444M 200/25mcg will be determined 0-24 hours (h) after dosing on Day 7 (primary endpoint). Secondary endpoints will include changes from baseline in QTcF, QT individual correction factor (QTci), QT duration corrected for heart rate by Bazett's formula (QTcB), and QT interval at each timepoint after 7 days dosing of fluticasone furoate/GW642444M 800/100mcg and single dose oral moxifloxacin (400mg) and changes from baseline in QTci, QTcB, and QT interval at each timepoint after 7 days dosing of fluticasone furoate/GW642444M 200/25mcg. Plasma concentrations (0-24h) and pharmacokinetic parameters of GW642444 and fluticasone furoate will also be derived.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 65 years of age inclusive.
* Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin ≤ 1.5xUpper limit of normal (ULN).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* A female subject is eligible to participate if she is of:

  • Non-childbearing potential defined as pre-menopausal females with tubal ligation or hysterectomy, and post-menopausal females. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods. All other female subjects must agree to use contraception until 4 months post-last dose.
* Body Mass Index (BMI) within 18.5-29.0 kilograms/metre2.
* Capable of giving written informed consent.
* Subjects who are current non-smokers, who have not used any tobacco products in the 6 month period preceding the screening visit.
* No significant abnormality on 12-lead ECG at screening.
* A 24 hour Holter ECG at screening which shows no abnormalities that could affect study data.
* Forced Expiratory Volume in 1 second (FEV1) ≥ 85% predicted at screening.
* Subjects who are able to use the inhaler satisfactorily.

Exclusion Criteria:

* Subject is deemed unsuitable for the study.
* A screening Holter ECG tracing that reveals clinically concerning arrhythmias
* A supine blood pressure that is persistently higher than 140/90 millimetres of mercury (mmHg) at screening.
* A supine mean heart rate outside the range 40-90 beats per minute (bpm) at screening.
* History or presence of any medically significant disease or disorder, in particular, a family history of QT prolongation, of early or sudden cardiac death or of early cardiovascular disease.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* The subject has any history of breathing problems in adult life.
* Subjects who have suffered an upper or lower respiratory tract infection within 4 weeks of the screening visit.
* Pregnant females.
* Lactating females.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for Human Immunodeficiency Virus (HIV) antibody.
* The subject has taken inhaled, intranasal or topical steroids less than 4 weeks before the screening visit.
* Positive carbon monoxide (CO) or alcohol breath test at screening or on admission to the Unit.
* Positive urine cotinine test at screening.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units for males or >14 units for females.
* The subject has participated in a clinical trial in the last 3 months.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days of the first dose.
* The subject has taken oral corticosteroids less than 8 weeks before the screening visit.
* History of sensitivity to any of the study medications.
* History of milk protein allergy.
* Where participation in the study would result in donation of blood or blood products in excess of 500 millilitres (mL) within a 90 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* Consumption of seville oranges, pommelos (members of the grapefruit family) or grapefruit juice from 7 days prior to the first dose of study medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2010-06-23 (Actual); Primary Completion 2011-01-04 (Actual); Study Completion 2011-01-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in QTcF interval at each timepoint on study Day 7 (average of at least 3 Holter ECG replicates per time point) for fluticasone furoate/GW642444M 200/25mcg as compared with time-matched placebo | Baseline and Day 7

SECONDARY OUTCOMES:
Change from baseline in QTcF interval at each timepoint on study Day 7 (average of at least 3 Holter ECG replicates per time point) for fluticasone furoate/GW642444M 800/100mcg as compared with time-matched placebo. | Baseline and Day 7
Change from baseline in QTci and QTcB interval at each timepoint on Study Day 7 (average of at least 3 Holter ECG replicates per time point) for fluticasone furoate/GW642444M 200/25mcg and 800/100mcg as compared with time-matched placebo | Baseline and Day 7
Change from baseline in QTcF interval at each timepoint on Study Day 7 (average of at least 3 Holter ECG replicates per time point) for moxifloxacin as compared with time-matched placebo. | Baseline and Day 7
Maximal change from baseline on Day 7 for QTcF, QTci and QTcB (for all treatments) | Baseline and Day 7
Change from baseline at each timepoint on Day 7 for other cardiac electrophysiological parameters: QT, QRS, RR, PR and ventricular rate (for all treatments) | Baseline and Day 7
Plasma concentrations of GW642444 and fluticasone furoate and derived pharmacokinetic parameters including maximum observed concentration(Cmax), time of occurence of Cmax (tmax), Area under the concentration-time curve over the dosing interval (AUC(0-τ)) | Study duration

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Kempsford R, Allen A, Kelly K, Saggu P, Crim C. A repeat-dose thorough QT study of inhaled fluticasone furoate/vilanterol combination in healthy subjects. Br J Clin Pharmacol. 2014 Mar;77(3):466-79. doi: 10.1111/bcp.12243. PMID 24093504
- See also: Results for study 102936 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/102936?search=study&search_terms=102936#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 102936 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 102936 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 102936 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 102936 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 102936 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 102936 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 102936 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register